CLINICAL TRIAL: NCT07171203
Title: Phase I Study of Neoadjuvant Therapy Imatinib Mesylate and Fampridine in KIT Mutant Gastrointestinal Stromal Tumor (GIST)
Brief Title: Neoadjuvant Imatinib and Fampridine in KIT Mutant Gastrointestinal Stromal Tumor
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Paul Fanta, Clinical professor, medical oncology, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 811484
Record Dates: First submitted 2025-09-05; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: imatinib; fampridine; 4-aminopyridine; gastrointestinal stromal tumor; phase 1 trial; KIT exon 11 mutant; voltage-gated potassium channel (VGKC) blocker
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Imatinib Mesylate; 4-Aminopyridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Imatinib plus Fampridine (Experimental): Imatinib in combination with fampridine at one of three dose levels (10 mg every other day, or 10 mg every day, or 10 mg twice a day) after a 7-day run-in period with imatinib monotherapy.
  Interventions: Drug: Imatinib; Drug: Fampridine

INTERVENTIONS:
Drug: Imatinib — Tyrosine kinase inhibitor. Imatinib will be dosed at 400 mg once a day. Dose can be reduced by 100 mg per dose reduction step if clinically indicated.
  Other Names: Imatinib mesylate; Gleevec
Drug: Fampridine — Voltage-gated potassium channel (VGKC) blocker. Fampridine will be dosed in a 3+3 design at 10 mg given either every 2 days, or every day, or twice a day.
  Other Names: Dalfampridine; Ampyra; Fampyra; 4-Aminopyridine

SUMMARY:
The goal of this clinical trial is to learn what dose of the drug fampridine can be given safely together with imatinib (Gleevec) in patients with gastrointestinal stromal tumor (GIST) with a DNA mutation in exon 11 of the KIT gene.

The main questions this study aims to answer are:

* What is the maximum dose of fampridine that can be given safely together with imatinib (Gleevec)?
* Is the combination of the two drugs efficacious against the tumor?

Participants will:

* Take the drugs before tumor surgery (neoadjuvant treatment) for at least 2 months with the option to continue for a longer period of time if treatment seems safe and effective.
* Visit the clinic at the scheduled appointments for checkups and tests.

DETAILED DESCRIPTION:
Gastrointestinal stromal tumor (GIST) is the most common form of sarcoma. Surgical resection is the current main form of treatment, however neoadjuvant medical therapies are also often necessary.

The majority of gastrointestinal stromal tumor (approximately 60-70%) are caused by gain-of-function mutations in the KIT oncogene. Since KIT is a tyrosine kinase, it is not surprising that four of five Food and Drug Administration (FDA)-approved therapies for this condition are tyrosine kinase inhibitors that target the KIT oncogene. Among these compounds, imatinib is considered the standard first line treatment. However, tumor response to tyrosine kinase inhibitors is suboptimal and more efficacious therapies are needed.

There are data that demonstrate lack of KIT protein expression in some KIT mutant gastrointestinal stromal tumor cells (cell not expressing KIT are referred to as KITnegative/low). Therefore, these cells do not have the cellular machinery that would allow them to respond to tyrosine kinase inhibitors.

The study investigators have discovered that the mRNA for the beta subunit of the voltage-gated potassium channels (VGKCs), Kvβ1.1, is expressed at high levels in KITnegative/low tumor cells. Previous studies have also shown that inhibition of the voltage-gated potassium channels (VGKCs) can inhibit cell proliferation and migration/invasion, as well as induce apoptosis in various cancer types. This led to the hypothesis that inhibitors of voltage-gated potassium channels (VGKCs) may have antitumor activity in KITnegative/low gastrointestinal stromal tumor cells.

A voltage-gated potassium channels inhibitor, fampridine, is FDA-approved for multiple sclerosis. The investigators hypothesize that voltage-gated potassium channels (VGKCs) blockade with fampridine may represent a novel strategy for treating KITnegative/low gastrointestinal stromal tumor. The investigators performed preclinical studies that suggest that the combination imatinib plus fampridine may lead to cell killing in an additive and/or synergistic manner in vitro. In addition, they showed that imatinib synergizes with fampridine to decrease tumor mass in vivo in a genetically engineered mouse model of GIST that carry KIT exon 11 Val-558 deletion.

Thus, the investigators aim to conduct this single site, prospective, open-label, non-randomized, single-arm phase 1 clinical trial in patients with KIT exon 11 mutant gastrointestinal stromal tumor to evaluate the safety and tolerability of the combination of imatinib plus fampridine in the neoadjuvant setting (before surgery) to establish the dose of fampridine that can be used in a future phase 2 trial.

The recommended phase 2 dose (RP2D) will be determined based on the rate of dose limiting toxicities (DLT) using the standard 3+3 phase 1 trial design with 3 dose levels.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent prior to any screening procedures
* Age ≥ 18 years
* Having been pathologically confirmed to have a KIT exon 11 mutant gastrointestinal stromal tumor assessed for KIT variant mutations by next generation sequencing
* Treatment naïve gastrointestinal stromal tumor
* Described as a primary localized or locally advance gastrointestinal stromal tumor in any location that would benefit from neoadjuvant therapy before tumor surgical resection
* Has measurable or evaluable disease per Response Evaluation Criteria in Solid Tumors v1.1.
* Has Eastern Cooperative Oncology Group Performance Status of 0-1
* Has adequate hematologic, hepatic, and renal function: Absolute Neutrophil Count ≥ 1.5 x 10^9/L; Hemoglobin ≥ 11 g/dL; Platelets ≥ 100 x 10^9/L; Serum total bilirubin < 2.0 x upper limit of normal; Aspartate aminotransferase and alanine aminotransferase ≤ 5 x upper limit of normal; Plasma creatinine phosphokinase < 1.5 x upper limit of normal; Serum creatinine ≤ 1.0 x upper limit of normal or calculated creatinine clearance ≥ 50ml/min based upon the Cockcroft-Gault Equation
* Life expectancy of ≥ 5 years
* Participants able to cause pregnancy agree to use an adequate method of contraception starting with the first dose of study therapy and for 120 days after the last dose

Exclusion Criteria:

* Unwilling or unable to comply with the protocol
* KIT exon 9, 13, 14, 17, or 18 mutant gastrointestinal stromal tumor by next generation sequencing.
* Non-KIT mutant gastrointestinal stromal tumor
* Newly diagnosed with metastatic gastrointestinal stromal tumor
* Have residual tumor following surgical debulking
* Have had major surgery within 4 weeks of initiation of study medication.
* Of childbearing potential
* Pregnant or nursing.
* Received imatinib monotherapy prior to the first dose of study treatment with imatinib plus fampridine and has demonstrated tumor shrinkage in computed tomography assessment images.
* Received fampridine prior to the first dose of study treatment with imatinib plus fampridine.
* Use of compounded fampridine or other forms of fampridine.
* Known brain metastases and any other progressive neurologic dysfunction should be excluded from this clinical trial because of their poor prognosis and because their progressive neurologic dysfunction would confound the evaluation of neurologic and other adverse events.
* Evidence of severe or uncontrolled systemic diseases (e.g., unstable, or uncompensated respiratory, cardiac [including life threatening arrhythmias] disease).
* Presence of cardiac impairment defined as:
* Prior history of cardiovascular disease including heart failure that meets New York Heart Association (NYHA) class III and IV definitions; OR
* History of myocardial infarction/active ischemic heart disease within one year of study entry; OR
* Uncontrolled dysrhythmias; OR
* Poorly controlled angina.
* Unresolved toxicity Common Terminology Criteria Adverse Events (CTCAE) Grade ≥ 2 from previous anti-cancer therapy.
* Allergy or sensitivity to fampridine or known allergies to aminopyridine products, which in the opinion of the investigator(s) suggests an increased potential for an adverse hypersensitivity to fampridine.
* Allergy to imatinib.
* Any chronic liver disease including, but not limited to cirrhosis, non-alcoholic steatohepatitis, alcohol-related liver disease, hemochromatosis, Wilson's disease, alpha-1 antitrypsin deficiency, hepatic, or biliary autoimmune disorders (i.e., primary biliary cholangitis, autoimmune hepatitis). Exception: Patients aged ≤ 65 years with non-alcoholic fatty liver disease detected by imaging are acceptable if adequate hepatic function as defined in the inclusion criteria is confirmed. Note: Patients aged > 65 years with non-alcoholic fatty liver disease are excluded from the study.
* Any evidence or history of hepatitis B and/or hepatitis C.
* Medical condition such as uncontrolled infection, uncontrolled diabetes mellitus or cardiac disease that, in the opinion of the investigator(s), would make this study unreasonably hazardous for the patient.
* Any other disease or clinically significant abnormality in laboratory parameters, including serious medical or psychiatric illness/condition, which in the judgment of the investigator(s) likely might compromise the safety of the participant or the integrity of the study, interfere with the participant participation in the trial, or compromise the trial objectives.
* History of seizures.
* Cannot swallow oral formulations of the medications or lack physical integrity of the upper gastrointestinal tract, or has known malabsorption syndromes. Note: imatinib tablets can be dissolved in water or apple juice if participants have difficulty swallowing.
* Have taken part in an experimental drug study within 4 weeks of initiating study treatment with imatinib plus fampridine
* Receiving other anti-neoplastic therapy (e.g., chemotherapy, targeted therapy, or radiotherapy) concurrently or within 4 weeks of starting study treatment with imatinib plus fampridine
* Receiving medications that inhibit the renal Organic Cation Transporter 2 (OCT2), such as cimetidine and quinidine, because of possible drug-drug interactions.
* Receiving medications known to be strong inhibitors or inducers of CYP3A4/5.
* Receiving medications known to be strong inhibitors or inducers of cytochrome CYP2E1 or medications metabolized by cytochrome CYP2B6 or CYP2C9/19 that have narrow therapeutic index and that cannot be discontinued before starting study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2030-07 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
Recommended phase 2 dose | 28 days
  Recommended phase 2 dose (RP2D) of imatinib plus fampridine determined by the dose-limiting toxicities and maximum tolerated dose via assessment of adverse events as defined by CTCAE version 5.0 during the first cycle (28 days) of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Fanta, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No